CLINICAL TRIAL: NCT05500144
Title: The Return to Work Experiences of People With Communication Disorders Post-stroke: a Qualitative Study
Brief Title: Return to Work With Post Stroke Communication Disorders
Acronym: ConQueSt
Status: Completed | Type: Observational
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1-017-22
Record Dates: First submitted 2022-06-16; First posted 2022-08-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- no intervention administered — Not applicable- no intervention administered

SUMMARY:
Approximately a quarter of stroke survivors are of working age, and it is well-known that disabilities caused by stroke can lead to difficulties returning to work. In addition to the economic cost, being out of the workplace due to disability has major psychosocial costs for the individual, causing reduced sense of purpose, quality of life, and standard of living. Communication problems (which can affect reading and writing, as well as producing and understanding speech) are not as visible as other stroke-related problems such as a weak arm or difficulties walking. However, they can cause major problems for returning to work because of the importance of communication across a vast range of work activities, for example as a means to engage with colleagues, to share information in order to solve problems and resolve conflicts, and as a means to ensure health and safety. There has been little research into the effects of communication problems on returning to work after a stroke, so the investigators want to explore this issue. Specifically, the investigators want to find out what helps and what hinders people with communication disorders following a stroke when they attempt to return to work; what information and support is most helpful to them; how this information and support should be given and by whom. The investigators aim to do this by interviewing people across NHS Grampian who have the experience of attempting to return to work with post-stroke communication problems. The investigators will then look at all the interviews together and find the common feelings or experiences that the participants mentioned. The findings will be written up and shared widely with professionals and with stroke survivors. The knowledge gained will help the investigators to plan a programme to help people with these problems to return to work.

ELIGIBILITY:
Inclusion Criteria:

Adults (aged 18 years of age and over) will be eligible if:

* they have had a stroke (excluding Transient Ischemic Attacks, or mini strokes) within the last 2 years
* they were in paid employment or actively seeking work at the time of their stroke
* they are attempting or have attempted (whether or not successfully) to return to paid employment since their stroke.

Exclusion Criteria:

Individuals will be excluded if:

* they lack the capacity to consent
* they are considered to have insufficient English language skills to be able to engage effectively in an interview, given that this is a small-scale study which will not have the resources to fund interpreter services
* they have a diagnosis of a learning disability, dementia or another comorbidity deemed to be as or more significant than the stroke in their experience of return to work.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (aged 18 years of age and over) who have post-stroke communication disorders, and who have attempted or are attempting to return to paid employment.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Experiences of returning or attempting to return to the workplace with post-stroke communication disorders | Through study completion, an average of 1 year
  Exploration of the experiences of people with post-stroke communication disorders returning or attempting to return to the workplace using semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Coutts, PhD, Principal Investigator — NHS Grampian
Locations (1):
- NHS Grampian, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT05500144/Prot_000.pdf